CLINICAL TRIAL: NCT06355921
Title: A Prospective Clinical Study on the Safety and Efficacy of Radiofrequency Ablation for the Treatment of Patients With Desmoid Tumors
Acronym: RFAdesmoid
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RFAdesmoid
Record Dates: First submitted 2024-03-29; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Desmoid Tumor; Desmoid Fibromatosis; Desmoid
MeSH Terms: conditions — Desmoid Tumors | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Desmoid (Experimental): Adult patients with desmoid tumors in the soft tissues of the extremities, trunk and paravertebral region of both sexes.In the study group, all patients after radiofrequency ablation of the tumor after 1 month will be evaluated using MRI and CT studies and, if solid components of the tumor are detected, repeated surgical treatment is performed followed by active monitoring after 1 month.
  In the absence of a solid component, the effect is estimated by the volume of the necrotic process and monitored in dynamics every 3 months.
  Interventions: Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: radiofrequency ablation — Anesthesia: Local (Novocaine, Lidocaine, Bupivacaine) Access: transcutaneous Navigation under CT control Cannulas are used: 22G 100 and 150 mm, the size of the electrode corresponds to the size of the cannula The starting power is 20W followed by steps of 10W every 2 minutes until the maximum power is reached, the maximum power is 60W.
  In order to prevent infectious complications, two-day antibiotic prophylaxis of Cefazolin (1g) is carried out 3 times a day In order to prevent skin burns with superficially located DFS, the skin is cooled during the procedure.

SUMMARY:
This is a prospective study on the safety and effectiveness of radiofrequency ablation in patients with desmoid tumors.

In the study group, all patients after radiofrequency ablation of the tumor after 1 month will be evaluated using MRI and CT studies and, if solid components of the tumor are detected, repeated surgical treatment is performed followed by active monitoring after 1 month.

In the absence of a solid component, the effect is estimated by the volume of the necrotic process and monitored in dynamics every 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically verified diagnosis of dermoid tumor
2. The presence of progressive, symptomatic or functionally significant DF.
3. Written Informed consent to participate in the study
4. Age from 18 to 75 years
5. The functional status of the patient according to the ECOG 0-2 scale
6. Normal renal function (estimated creatinine clearance 60 ml/min);
7. Normal level of bilirubin and liver enzymes (AST, ALT - no more than 3 norms);
8. Left ventricular ejection fraction > 55%
9. Satisfactory bone marrow function (hemoglobin level 9 g/dl, neutrophil count 1.5 thousand/ml, platelet count < 100 thousand/ml);

Exclusion Criteria:

1. The inability to obtain informed consent to participate in the study
2. Synchronous or metachronous cancer
3. Clinically significant diseases of the cardiovascular system
4. Clinically significant CNS diseases
5. Previous grade 2 polyneuropathy and above
6. Current infection or other severe or systemic disease that increases the risk of complications of therapy
7. Pregnancy, lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of safety assessment. | The effectiveness of treatment is monitored 1 month after treatment, then every 3 months for 2 years, every 6 months from 2 to 3 years from the moment of therapy
  Adverse Event Assessment and Serious Adverse Event Assessment according to CTCAE 5.0

SECONDARY OUTCOMES:
Overall Response Rate | The effectiveness of treatment is monitored 1 month after treatment, then every 3 months for 2 years, every 6 months from 2 to 3 years from the moment of therapy
  Proportion of patients who have a partial or complete response to therapy
Duration of responce | 3 years
  The time from randomization to disease progression or death for patients who achieve complete or partial alleviation
Comparison of tumor necrosis based on MRI/CT | The effectiveness of treatment is monitored 1 month after treatment, then every 3 months for 2 years, every 6 months from 2 to 3 years from the moment of therapy
  Proportion of tumor necrosis after therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budgetary Institution "N.N. Blokhin National Medical Research Center of Oncology" оf the Ministry of Health of the Russian Federation (N.N. Blokhin NMRCO), Moscow, Moscow Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
URL: https://www.ronc.ru/